CLINICAL TRIAL: NCT07386847
Title: Real-world Treatment Patterns and Effectiveness Among Patients With Locally Advanced or Metastatic Urothelial Carcinoma (la/mUC)
Brief Title: A Real-world Study of the First Treatment and Outcomes of Patients With Advanced or Metastatic Bladder Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C5701010
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Urothelial Carcinoma; Urothelial Cancer; Urothelial Carcinoma; Locally Advanced or Metastatic Urothelial Carcinoma
Keywords: Metastatic Urothelial Carcinoma; Locally Advanced or Metastatic Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- la/mUC: Patients with Locally Advanced or Metastatic Urothelial Carcinoma (la/mUC) who received first line treatment.

SUMMARY:
Bladder cancer (urothelial carcinoma) is a disease where cells in the bladder grow out of control. The bladder is an organ in the lower part of the body that stores urine. When someone has bladder cancer, abnormal cells form in the bladder and can spread to other parts of the body if not treated. Bladder cancer that has spread outside the bladder is called advanced or metastatic bladder cancer.

The purpose of this study is to examine how long it takes for adults with advanced or metastatic bladder cancer to experience worsening of their disease following their first treatment . The researchers will also describe which medicines these patients use as their first treatment for the disease.

This is a real-world study, not a clinical study. This means that researchers will look at what happens when patients receive the treatments prescribed by their own doctor as part of their usual healthcare treatment. In this study, researchers will use information from cancer clinics (Flatiron Health electronic health records). The study will include patients' information from the database who:

* Were identified to have advanced or metastatic bladder cancer.
* Started their first treatment after 01 Apr 2023.
* Were 18 years of age or older when they were diagnosed with advanced disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older) diagnosed with locally advanced or metastatic urothelial carcinoma (la/mUC) in the Flatiron Health database.
* Started first line systemic treatment for la/mUC during the study period.
* Received care in the United States, as the study is U.S.-based.
* Has sufficient available real-world data to assess treatment patterns and outcomes (e.g., treatment dates, follow-up, response/survival information).

Exclusion Criteria:

* Histology other than transitional cell (urothelial) carcinoma.
* Primary site of disease other than bladder, renal pelvis, ureter, or urethra
* Clinical trial participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients in the United States diagnosed with locally advanced or metastatic urothelial carcinoma (la/mUC) who initiated first line systemic treatment in the Flatiron Health database after 04/01/2023.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Real-world Progression Free Survival (rwPFS) | Up to 2 Years
  Time from initiation of first line treatment for la/mUC to the earliest of disease progression or death, based on real-world data sources.

SECONDARY OUTCOMES:
Real-world Overall Tumor Response (rwOTR) | Up to 2 Years
  Proportion of patients achieving tumor response (e.g., complete or partial response) based on real-world oncology data.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.